CLINICAL TRIAL: NCT04509375
Title: Comparison of Results of Near-Infrared Spectroscopy and Cranial Doppler Measurements in Premature Newborns With Anemia
Brief Title: Near-Infrared Spectroscopy and Cranial Doppler in Premature Newborns With Anemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, Associate Professor of Neonatology, Hacettepe University
Other Study IDs: KA-19030
Record Dates: First submitted 2020-08-04; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Anemia of Prematurity
Keywords: Newborn; Anemia; Near-infrared spectroscopy; Cranial doppler ultrasonography
MeSH Terms: conditions — Anemia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Premature babies in the first 28 postnatal days of life, with less than 32 gestational weeks or less than 1500 grams of birth weight, with documented anemia by current accepted transfusion guidelines of Turkish Neonatal Society
  Interventions: Device: Cranial Doppler Ultrasonography; Device: Near-Infrared Spectroscopy

INTERVENTIONS:
Device: Cranial Doppler Ultrasonography — Before and after the transfusions, flow measurements of middle cerebral arteries will be obtained.
Device: Near-Infrared Spectroscopy — Before, during and after the transfusions, regional cerebral oxygen saturation measurements will be obtained.

SUMMARY:
It is aimed in this study to examine the changes in brain blood supply and oxygenation in neonatal premature babies who have anemia and who underwent erythrocyte suspension transfusion in the light of original guidelines by means of obtaining measurements with the help of cranial doppler ultrasonography and near-infrared spectroscopy.

DETAILED DESCRIPTION:
Anemia in newborn babies is defined as the mean of hemoglobin values according to postnatal age is below 2 standard deviations. Disruption in tissue perfusion and oxygenation, hyperdynamic cardiac failure, increase in need of oxygen, increase in respiratory effort, inability to be separated from mechanical ventilation, failure to thrive, paleness, increase in frequency of morbidities of prematurity (necrotizing enterocolitis, retinopathy of prematurity, intraventricular hemorrhage, etc.) may be seen as a result of progressive anemia. When critical hemoglobin values are reached in premature newborn babies with concomitant disruption of tissue oxygenation, transfusion is performed with erythrocyte suspensions. The main goal here is to correct impaired tissue oxygenation, provide perfusion in sufficient quantity, and prevent anemia-related morbidities. Although frequently applied, there is no consensus in our country and in the world regarding threshold hemoglobin values and supporting parameters for transfusions. As a result, there are no guidelines prepared for newborns based on evidence with clearly defined borders and accepted by everyone. Many countries and centers implement different transfusion protocols based on their experience. Given the risk of oxygen radical damage and associated diseases as a result of erythrocyte transfusions (infections, bone marrow suppression, necrotizing enterocolitis, retinopathy of prematurity, etc.), there is a need to develop new methods for taking and supporting transfusion decision, and to prepare more objective and more accepted guidelines. The origin of our study is the subsequent protective compensation mechanisms after deterioration in brain oxygenation due to symptomatic anemia in premature newborn babies. For these reasons, it is aimed to examine the changes in brain blood supply and oxygenation in neonatal premature babies who have anemia and who underwent erythrocyte suspension transfusion in the light of original guidelines by means of obtaining measurements with the help of cranial doppler ultrasonography and near-infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

Premature babies less than 32 gestational weeks or less than 1500 grams of birth weight and Documented anemia in postnatal 28 days according to Turkish Neonatal Society guidelines

Exclusion Criteria:

Babies older than postnatal 28 days Major congenital anomalies Chromosomal anomalies Inborn errors of metabolism Hypoxic ischemic encephalopathy Disseminated intravascular coagulation Unstable hemodynamic status Severe neonatal sepsis Patients who are not volunteered to participate

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature babies in the first 28 postnatal days of life, with less than 32 gestational weeks or less than 1500 grams of birth weight, with documented anemia by current accepted transfusion guidelines of Turkish Neonatal Society
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-06-23 (Estimated); Study Completion 2021-06-23 (Estimated)

PRIMARY OUTCOMES:
Gradual improvement in middle cerebral artery flow patterns obtained by cranial doppler ultrasound imaging | Cranial doppler ultrasonography measurements will be obtained immediately before and 4 hours after the trasfusions.
  After a critical point, the cerebral oxygenation will be compromised due to anemia in spite of normal compensation mechanisms of cerebral vasculature. Erythrocyte suspension transfusion will help to normalize altered cerebral blood flow. It is hypothesized that these changes can be detected by cranial doppler ultrasonography as follows: Middle cerebral artery peak systolic velocity and flow volume will be increased before transfusion, possibly indicating the need of intervention. Four hours after transfusion, middle cerebral artery peak systolic velocity and flow volume will gradually fall and reach eventually a steady normal state. This in turn may also serve to better understand the effectiveness of the transfusion.
Gradual improvement in regional cerebral oxygen saturation measures obtained by near-infrared spectroscopy (NIRS) | NIRS measurements will be obtained 4 hours before, 2 hours during, and 4 hours after the trasfusions.
  After a critical point, the cerebral oxygenation will be compromised due to anemia in spite of normal compensation mechanisms of cerebral vasculature. Erythrocyte suspension transfusion will help to normalize altered cerebral blood flow. It is hypothesized that these changes can be measured by near-infrared spectroscopy (NIRS) as follows: Regional cerebral oxygen saturations (cSO2) will be low before transfusion, possibly indicating the need of intervention. During transfusion time of 2 hours, cSO2 will rise gradually and reach eventually a steady normal state in 4 hours after transfusion. This in turn may also serve to better understand the effectiveness of the transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Aykanat, Principal Investigator — Hacettepe University; Ercan Ayaz, Principal Investigator — Hacettepe University; Nursun Özcan, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aranha CA, Lederman HM, Segre CA. Color Doppler evaluation of the influence of type of delivery, sex, postnatal age and time post feeding on full term healthy newborns cerebral blood flow. Arq Neuropsiquiatr. 2009 Jun;67(2B):463-73. doi: 10.1590/s0004-282x2009000300017. PMID 19623445
- [Background] Sood BG, McLaughlin K, Cortez J. Near-infrared spectroscopy: applications in neonates. Semin Fetal Neonatal Med. 2015 Jun;20(3):164-72. doi: 10.1016/j.siny.2015.03.008. Epub 2015 Apr 29. PMID 25934116